CLINICAL TRIAL: NCT06692504
Title: Real-life Epidemiology of Adverse Drug Events in Patients on Oral Anticoagulation in the Emergency Department Setting
Brief Title: Adverse Drug Events in Patients on Oral Anticoagulation in the Emergency Department
Acronym: ADEOA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/920
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Hemorrhage; Thrombosis; Anticoagulant Therapy; Traumatic Hemorrhage
Keywords: anticoagulant therapy; oral anticoagulant; emergency department; emergency medicine; hemorrhage; Traumatic hemorrhage; Spontaneous hemorrhage; Asymptomatic overdose; Thrombosis; epidemiology; mortality
MeSH Terms: conditions — Hemorrhage; Thrombosis; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Oral anticoagulant therapy: anti-vitamin K or direct oral anticoagulants therapy
- No oral anticoagulant therapy: no anti-vitamin K or direct oral anticoagulants therapy

SUMMARY:
Rationale:

According to the latest National Survey on Care-Related Adverse Events, anticoagulants, including vitamin K antagonists (VKAs), rank first among medications responsible for serious iatrogenic accidents (37% in 2004, 31% in 2009). The EMIR study (2007) showed that VKAs were the leading cause of hospitalization for adverse effects (12.3%), with approximately 5,000 fatal hemorrhage-related accidents annually. Treatment and prevention of thromboembolic events represent a major public health challenge due to increased mortality, severity of functional sequelae, growing number of patients requiring treatment, and medical, social, and economic consequences. In 2013, an estimated 3.12 million patients received anticoagulation (4-5% of the French population). Several types of adverse events under oral anticoagulation appear to have high incidence in emergency settings: traumatic hemorrhage, spontaneous hemorrhage, asymptomatic overdose, and thrombosis. Different variables are associated with these events in patients admitted to emergency departments under oral anticoagulant treatment, but few studies have been conducted in real-world settings with large patient samples.

Hypothesis:

Iatrogenic events have a high incidence in patients admitted to emergency departments under oral anticoagulants and are a factor in early and late morbidity and mortality.

Primary Objective:

To describe the characteristics of patients admitted to the emergency department on oral anticoagulant therapy, with a particular focus on characterizing those presenting with Adverse Drug Events (ADEOA).

Study Design:

* Type: Observational, descriptive study
* Duration: 36 months total (24 months for data collection, 12 months for analysis)
* Sample Size: Estimated 2,080 patients (approximately 20 patients/week over 2 years)

Inclusion Criteria:

* Age ≥18 years
* Admission to adult emergency department
* Study period: January 1, 2018 to December 31, 2019
* Current oral anticoagulation therapy with:

  * Acenocoumarol (Sintrom®/Minisintrom®)
  * Apixaban (Eliquis®)
  * Dabigatran (Pradaxa®)
  * Fluindione (Previscan®)
  * Rivaroxaban (Xarelto®)
  * Warfarin (Coumadine®)

Exclusion Criterion:

- Discontinuation of anticoagulant therapy for more than 24 hours

Primary Outcome Measures:

1. Description of oral anticoagulant groups based on medication type
2. Characterization of Adverse Drug Events in Patients on Oral Anticoagulation in the Emergency Department (ADEOA):

   1. Presence of ADEOA:

      * Traumatic hemorrhage: acute bleeding following recent trauma
      * Spontaneous hemorrhage: acute bleeding unrelated to recent trauma
      * Asymptomatic overdose: INR >3 for vitamin K antagonist patients
      * Thrombosis: new arterial or venous thrombosis despite ongoing anticoagulation
   2. Absence of ADEOA

Secondary Outcome Measures:

1. Assessment of adherence to oral anticoagulant prescribing guidelines
2. Identification of etiological factors for anticoagulation-related adverse events
3. Identification of early morbidity and mortality risk factors
4. Evaluation of medical-economic impact of adverse events and cost-effectiveness analysis of adverse events
5. Quality of life assessment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Admission to adult emergency department of Besançon University Hospital
* Study period: January 1, 2018 to December 31, 2019
* Current oral anticoagulation therapy with:

  * Acenocoumarol
  * Apixaban
  * Dabigatran
  * Fluindione
  * Rivaroxaban
  * Warfarin

Exclusion Criterion:

- Discontinuation of anticoagulant therapy for more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients on oral anticoagulation therapy admitted to the emergency department
Sampling Method: Probability Sample
Enrollment: 2080 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Description of oral anticoagulant groups based on medication type | 1 day

SECONDARY OUTCOMES:
Characterization of Iatrogenic Events Related to Oral Anticoagulants (ADEOA) | 1 day
  * Traumatic hemorrhage: acute bleeding following recent trauma
  * Spontaneous hemorrhage: acute bleeding unrelated to recent trauma
  * Asymptomatic overdose: INR >3 for vitamin K antagonist patients
  * Thrombosis: new arterial or venous thrombosis despite ongoing anticoagulation
Assessment of adherence to oral anticoagulant prescribing guidelines | 1 day
Identification of etiological factors for anticoagulation-related adverse events | 1 day
Identification of early morbidity and mortality risk factors | 1 year
Evaluation of medical-economic impact of adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric MAUNY, MD, PhD, Study Chair — CHU Besançon; Marc PUYRAVEAU, MSc, Study Chair — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided